CLINICAL TRIAL: NCT05764486
Title: A Study About the Operation Efficacy and the Early Stage Safety of Heavy Ion Beam Treatment System in Solid Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-02-013C
Record Dates: First submitted 2023-02-24; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment plan (Other): Treatment plan performed by Hitachi's Heavy Ion Beam Therapy System HyBEAT will be designed to suit the particular needs of each subject and the course of treatment will differ for each subject depending on the type of tumor, varying from 1 day to 4 weeks. All subjects will be monitored for 12 weeks after receiving the last treatment.
  Interventions: Device: Hitachi's Heavy Ion Beam Therapy System HyBEAT

INTERVENTIONS:
Device: Hitachi's Heavy Ion Beam Therapy System HyBEAT — treating patients with solid tumor

SUMMARY:
The main purpose of this study is to investigate the safety of Hitachi's Heavy Ion Beam Therapy System HyBEAT for treating patients with solid tumor in Taipei Veterans General Hospital, including patients early-stage adverse reactions and the efficacy on tumors, as well as to assess the operation efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 20 years of age inclusive, male or female
2. Diagnosed with one of the following cancer: head and neck cancer, lung cancer, liver cancer, prostate cancer, osteosarcoma or bone and soft-tissue tumours
3. Having a lesion of less than 12cm
4. Having no metastasis at distant organ sites
5. Having a life expectancy of more than 12 weeks or longer
6. ECOG Performance Status (ECOG PS): 0, 1 or 2
7. Maintain the function of major organs and satisfy the following criteria: WBC≥3,000 / mm3 , Plt

   ≥75,000 / mm3 (assuming no serious bleeding tendency below 100,000), Hb≥9.5 g / dl
8. Able to maintain body position during irradiation
9. Based on his/her free will, agree to participate in the clinical study and sign and date the informed consent form after understanding the clinical study.

Exclusion Criteria:

1. Weigh more than or equal to 135kg
2. Subjects need chemotherapy or immunotherapy as concomitant treatment
3. Have received radiotherapy on the area planned to be irradiated
4. Have received local treatment that might potentially affect endpoint evaluation, 4 weeks prior to the screening process (for instance TACE etc.)
5. Have been treated with targeted therapy, chemotherapy or immunotherapy 4 weeks prior to the screening process
6. Participated in other clinical studies within 12 weeks before screening (studies using questionnaire are exemption)
7. Subjects contraindicated in using radiotherapy
8. Wearing electronic devices, for example implantable cardiac pacemakers, implantable defibrillators, cerebrospinal stimulators, artificial hearts and cochlear implants, where the function and activity may be affected by radiation
9. Have been diagnosed with another active, uncontrolled cancer
10. Subjects whose irradiated area has active or persistent infectious disease
11. Has autoimmune diseases or connective tissue diseases
12. Subjects with other serious complications
13. Pregnant or currently breastfeeding
14. Planning to give birth or unable to take contraception during the screening and treatment period, as well as within 52 weeks after receiving the last treatment, regardless of gender.
15. Subjects who are judged by the investigators as unsuitable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Adverse event | up to 12 weeks
  The adverse reactions and the severity of all subjects in the early stage will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Li, Lan, Principal Investigator — Doctor
Locations (1):
- Cancer Center, Taipei Veterans General Hospital, Taipei, Taiwan